CLINICAL TRIAL: NCT00044694
Title: A Phase 2, Randomized, Triple-Blind, Placebo-Controlled, Short-Term, Dose-Response Study to Examine the Effect on Glucose Control and Safety and Tolerability of AC2993 Given Two Times a Day in Subjects With Type 2 Diabetes Mellitus
Brief Title: Evaluation of the Effect on Glucose Control and the Safety and Tolerability of AC2993 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2993-116
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo 0.01 mL (Placebo Comparator): 2 week placebo lead-in followed by Placebo 0.01 mL
  Interventions: Drug: Placebo 0.01 mL
- Placebo 0.02 mL (Placebo Comparator): 2 week placebo lead-in followed by Placebo 0.02 mL
  Interventions: Drug: Placebo 0.02 mL
- Placebo 0.03 mL (Placebo Comparator): 2 week placebo lead-in followed by Placebo 0.03 mL
  Interventions: Drug: Placebo 0.03 mL
- Placebo 0.04 mL (Placebo Comparator): 2 week placebo lead-in followed by Placebo 0.04 mL
  Interventions: Drug: Placebo 0.04 mL
- AC2993 2.5 mcg (Experimental): 2 week placebo lead-in (0.01 mL) followed by AC2993 2.5 mcg; 0.01 mL
  Interventions: Drug: AC2993 2.5 mcg
- AC2993 5.0 mcg (Experimental): 2 week placebo lead-in followed by AC2993 5.0 mcg; 0.01 mL
  Interventions: Drug: AC2993 5.0 mcg
- AC2993 7.5 mcg (Experimental): 2 week placebo lead-in followed by AC2993 7.5 mcg; 0.03 mL
  Interventions: Drug: AC2993 7.5 mcg
- AC2993 10.0 mcg (Experimental): 2 week placebo lead-in period followed by AC2993 10.0 mcg; 0.04 mL
  Interventions: Drug: AC2993 10.0 mcg

INTERVENTIONS:
Drug: Placebo 0.01 mL — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of Placebo 0.01 mL subcutaneously injected twice daily
  Arms: Placebo 0.01 mL
Drug: Placebo 0.02 mL — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of Placebo 0.02 mL subcutaneously injected twice daily
  Arms: Placebo 0.02 mL
Drug: Placebo 0.03 mL — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of Placebo 0.03 mL subcutaneously injected twice daily
  Arms: Placebo 0.03 mL
Drug: Placebo 0.04 mL — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of Placebo 0.04 mL subcutaneously injected twice daily
  Arms: Placebo 0.04 mL
Drug: AC2993 2.5 mcg — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of AC2993 2.5 mcg (0.01 mL) subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 2.5 mcg
Drug: AC2993 5.0 mcg — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of AC2993 5.0 mcg (0.02 mL) subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 5.0 mcg
Drug: AC2993 7.5 mcg — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of AC2993 7.5 mcg (0.03 mL) subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 7.5 mcg
Drug: AC2993 10.0 mcg — 2-week placebo lead-in period (0.01 mL) followed by 4 weeks of AC2993 10.0 mcg (0.04 mL) subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 10.0 mcg

SUMMARY:
This is a multicenter, randomized, blinded, placebo-controlled, short-term, dose-response study to examine the effects on glucose control of AC2993 as compared to placebo in patients with type 2 diabetes. Patients will be individuals with type 2 diabetes treated with metformin for at least 3 months prior to screening. Patients whose diabetes management consists of diet and exercise will also be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Treated with diet and exercise alone or with metformin for at least 3 months prior to screening
* BMI 27-45 kg/m^2
* HbA1c between 7.0 % and 8.0 %

Exclusion Criteria:

* Treated with other oral anti-diabetic agents other than metformin within 3 months of screening
* Patients previously treated with AC2993
* Patients presently treated with insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2002-08; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Day 28 | Baseline (Day 1) to Day 28
  Change in HbA1c from Baseline (Day 1) to study termination (Day 28)

SECONDARY OUTCOMES:
Change in HbA1c from Baseline to Day 14 | Baseline, Day 14
  Change in HbA1c from Baseline (Day 1) to Day 14
Change in fasting plasma glucose from Baseline to Day 14 and to Day 28 | Baseline, Day 14, Day28
  Change in fasting plasma glucose from Baseline (Day 1) to Day 14 and to study termination (Day 28)
Change in serum fructosamine from Baseline (Day 1) to Day 14 and to Day 28 | Baseline, Day 14, Day 28
  Change in serum fructosamine from baseline (Day 1) to Visit 4 (Day 14) and to study termination (Day 28)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Innovative Clinical Trials, Birmingham, Alabama
  - Healthsouth Clinical Research, Birmingham, Alabama
  - Endocrinology Clinic of O.C., Anaheim, California
  - Pioneer Medical Group, Bellflower, California
  - International Clinical Research Network, Chula Vista, California
  - Bautista Research and Medical Clinic, Fresno, California
  - Whittier Institute for Diabetes, La Jolla, California
  - Richard Cherlin, M.D., Los Gatos, California
  - Dr. Martinez Medical Clinic, Moreno Valley, California
  - Anshutz Outpatient Pavilion, Aurora, Colorado
  - Diagnostic Clinic, Clearwater, Florida
  - Radiant Research-Gainsville, Gainsville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Radiant Research-Pinellas Park, Pinellas Park, Florida
  - Clinical Research Group of North Georgia, Blairsville, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Radiant Research-Honolulu, Honolulu, Hawaii
  - Radiant Research-Boise, Boise, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Northshore Medical Research, LLC, Covington, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Melvin Kramer, MD, Concord, Massachusetts
  - Radiant Research-Edina, Edina, Minnesota
  - Mississippi Medical Research, LLC, Gulfport, Mississippi
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Innovative Health Research, Las Vegas, Nevada
  - Carolina Advanced Research, Cary, North Carolina
  - Fallen Timbers Internal Medicine, LLC, Maumee, Ohio
  - Millenium Research, Benbrook, Texas
  - Healthsouth Clinical Research, DeSoto, Texas
  - Baylor College of Medicine/Clinical Studies Unit, Houston, Texas
  - Diabetes Center of the Southwest, Midland, Texas
  - Utah Diabetes Center at the University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Nelson P, Poon T, Guan X, Schnabel C, Wintle M, Fineman M. The incretin mimetic exenatide as a monotherapy in patients with type 2 diabetes. Diabetes Technol Ther. 2007 Aug;9(4):317-26. doi: 10.1089/dia.2006.0024. PMID 17705687